CLINICAL TRIAL: NCT03579511
Title: Delivery of Fetal Head During Cesarean Section; Acceptability and Learning Curve of External Pop Out as a New Technique for Lower Uterine Segment Support; A Cross- Sectional Study
Brief Title: Learning Curve of External Pop Out as a New Technique for Lower Uterine Segment Support
Acronym: EPO
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: EPOLC
Record Dates: First submitted 2018-06-26; First posted 2018-07-06 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: External Pop-out — The original techniques of fetal head extraction entail the introduction of the obstetricians' hands or other instruments into the LUS. This puts the LUS at risk of damage and incision extensions with its consequences of increased blood loss, increased operative time,infection adhesions and blood transfusion.To the available, the generated good quality evidence bases practice in CS is anticipated to decrease such morbidities

SUMMARY:
Cesarean section represent the most significant operative intervention in all of obstetrics, its development and application have saved lives of countless mothers and infants. the frequency with which its carried out continues to rise and has in many hospitals and health regions reached rates in excess of 30%(

ELIGIBILITY:
Inclusion Criteria:

1. Singleton term pregnancy
2. Cephalic presentation
3. Women who will accept to participate in the study

Exclusion Criteria:

1. Non-cephalic presentation
2. Congenital fetal anomalies
3. Multiple pregnancy
4. Preterm caesarean < 37 weeks
5. Cases with marked adhesions obscuring the lower uterine segment thickness

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: B. Eligible women who will present to the hospital and fulfill the inclusion criteria during the study period will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
The number of cesarean sections that are required for the obstetrician to reach turning point . | 1 month
  the number needed to achieve a good learning curve

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt